CLINICAL TRIAL: NCT00560313
Title: A Phase 2, Multi-Center, Open-label Study of the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine When Administered at a 0, 2, 6-Month Schedule and of a Single Dose of Novartis Meningococcal ACWY Conjugate Vaccine in Healthy At-risk Adults 18-50 Years of Age
Brief Title: Safety, Tolerability and Immunogenicity of Three Doses of Novartis Meningococcal B Vaccine When Administered to Healthy At-risk Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: V72P4; 2007-001563-29
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal disease; prevention; vaccination
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4CMenB (Experimental)
  Interventions: Biological: 4CMenB
- MenACWY CRM (Experimental)
  Interventions: Biological: Men ACWY CRM

INTERVENTIONS:
Biological: Men ACWY CRM — A single dose of a 0.5 mL injectable solution
  Arms: MenACWY CRM
Biological: 4CMenB — All subjects received the study vaccine following a 0,2,6 vaccination schedule. Pre-filled syringe, administered by intramuscular injection into the deltoid area of the non dominant arm.
  Arms: 4CMenB

SUMMARY:
This study is aimed to evaluate safety, tolerability and immunogenicity of three doses of Novartis 4CMenB and of one dose of Novartis Meningococcal ACWY vaccine when administered to healthy at-risk adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults,18 through 50 years of age, who were or might be routinely exposed to N. meningitidis cultures

Exclusion Criteria:

* Previous ascertained or suspected disease caused by N. meningitidis;
* Pregnancy or breastfeeding;
* History of any anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component;
* Any present or suspected serious acute or chronic disease
* Known or suspected autoimmune disease or impairment /alteration of immune function

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2007-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Director — Novartis Vaccines
Locations (1):
- Azienda USL 7 of Siena, Siena, Italy

REFERENCES:
- [Result] Kimura A, Toneatto D, Kleinschmidt A, Wang H, Dull P. Immunogenicity and safety of a multicomponent meningococcal serogroup B vaccine and a quadrivalent meningococcal CRM197 conjugate vaccine against serogroups A, C, W-135, and Y in adults who are at increased risk for occupational exposure to meningococcal isolates. Clin Vaccine Immunol. 2011 Mar;18(3):483-6. doi: 10.1128/CVI.00304-10. Epub 2010 Dec 22. PMID 21177912
- [Derived] Bartolini E, Borgogni E, Bruttini M, Muzzi A, Giuliani M, Iozzi S, Petracca R, Martinelli M, Bonacci S, Marchi S, Brettoni C, Donati C, Torricelli G, Guidotti S, Domina M, Beninati C, Teti G, Felici F, Rappuoli R, Castellino F, Del Giudice G, Masignani V, Pizza M, Maione D. Immunological fingerprint of 4CMenB recombinant antigens via protein microarray reveals key immunosignatures correlating with bactericidal activity. Nat Commun. 2020 Oct 5;11(1):4994. doi: 10.1038/s41467-020-18791-0. PMID 33020485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one site in Italy and one site in Germany.
Pre-assignment Details: Approximately 250 adults were planned to be enrolled in this study but only a total of 54 subjects were enrolled after the screening for the inclusion and exclusion criteria.
Groups:
- 4CMenB: All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB
Period: Overall Study
Arm/Group | 4CMenB
Started | 54
Completed | 48
Not Completed | 6
Not completed — Adverse Events or Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | 4CMenB
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer of the Meningococcal B Vaccine Against the Different Strains at One Month After First, Second and Third Vaccination.
Description: Geometric mean titers(GMT) and the respective confidence intervals measured after each vaccination against the three different meningococcal strains.
Time Frame: One month after vaccinations
Population: The analysis was done on the per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 4CMenB (44/76-SL): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. Response was measured against (44/76-SL) strain
- 4CMenB (5/99): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. Response was measured against the (5/99)strain
- 4CMen B (NZ98/254): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. Response was measured against the (NZ98/254)strain.
Arm/Group | 4CMenB (44/76-SL) | 4CMenB (5/99) | 4CMen B (NZ98/254)
Number analyzed (Participants) | 46 | 46 | 46
titer
  Baseline titer | 2.5 [1.7 to 3.5] | 2.3 [1.6 to 3.2] | 1.8 [1.3 to 2.6]
  Post dose 1 titer (N=25) | 33 [15 to 72] | 29 [14 to 60] | 23 [11 to 49]
  Post dose 2 titer | 93 [71 to 121] | 144 [108 to 193] | 32 [21 to 48]
  Before dose 3 titer(N=24) | 26 [15 to 47] | 37 [26 to 53] | 9.4 [4.1 to 21]
  Post dose 3 titer (N=39) | 95 [68 to 131] | 269 [205 to 354] | 30 [18 to 50]

2. Primary Outcome: Percentages of Participants With Serum Bactericidal Activity of the Meningococcal B Vaccine Against Different Strains at One Month After First, Second and Third Vaccination.
Description: Percentage of participants with serum bactericidal activity (SBA) of the Meningococcal ACWY vaccine at one month after vaccination against A, C, W-135 and Y strains. Bactericidal activity (% ≥ 1:4, i.e., percentage of subjects with BCA titer ≥ 1:4; % ≥ 1:8, i.e. percentage of subjects with BCA titer ≥ 1:8) against a panel of genetically distinct meningococcal B strains:
  * prior to the first vaccination
  * 30 days following the first, second, prior to the third and 30 days after the third vaccination
Time Frame: One month after vaccinations
Population: The analysis was done on the per protocol population.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- 4CMenB (5/99): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. Response was measured against the (5/99) strain
- 4CMen B (NZ98/254): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. Response was measured against the (NZ98/254) strain.
Arm/Group | 4CMenB (44/76-SL) | 4CMenB (5/99) | 4CMen B (NZ98/254)
Number analyzed (Participants) | 46 | 46 | 46
percentage
  titer ≥4 (Baseline) | 37 [23 to 52] | 37 [23 to 52] | 22 [11 to 36]
  titer ≥4 (Post dose 1) N=25 | 84 [64 to 95] | 88 [69 to 97] | 80 [59 to 93]
  titer ≥4 (Post dose 2) | 100 [92 to 100] | 100 [92 to 100] | 91 [79 to 98]
  titer ≥4 (Before dose 3) N=24 | 96 [79 to 100] | 100 [86 to 100] | 67 [45 to 84]
  titer ≥4 (Post dose 3) N=39 | 97 [87 to 100] | 100 [91 to 100] | 92 [79 to 98]
  titer ≥8 (Baseline) | 26 [14 to 41] | 15 [6 to 29] | 15 [6 to 29]
  titer ≥8 (Post dose 1) N=25 | 80 [59 to 93] | 76 [55 to 91] | 72 [51 to 88]
  titer ≥8 (Post dose 2) | 100 [92 to 100] | 100 [92 to 100] | 83 [69 to 92]
  titer ≥8 (Before dose 3) N=24 | 75 [53 to 90] | 100 [86 to 100] | 54 [33 to 74]
  titer ≥8 (Post dose 3) N=39 | 97 [87 to 100] | 100 [91 to 100] | 77 [61 to 89]
  ≥4 fold increase (Post dose 1) N=25 | 80 [59 to 93] | 64 [43 to 82] | 68 [46 to 85]
  ≥4 fold increase (Post dose 2) | 100 [92 to 100] | 100 [92 to 100] | 78 [64 to 89]
  ≥4 fold increase (Before dose 3) N=24 | 71 [49 to 87] | 75 [53 to 90] | 46 [26 to 67]
  ≥4 fold increase (Post dose 3) N=39 | 92 [79 to 98] | 100 [91 to 100] | 69 [52 to 83]

3. Primary Outcome: Geometric Mean Titer (GMT) of the Meningococcal ACWY Vaccine at One Month After Vaccination.
Description: Geometric mean titer (GMT) of the Meningococcal ACWY Vaccine at One Month After the Immunization against the A, C, W-135 and Y strains.
Time Frame: One month after vaccinations
Population: The analysis was done on the per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- MenACWY-CRM (A); MenACWY-CRM (C); MenACWY-CRM (W-135); MenACWY-CRM (Y): 1 month postvaccination with quadrivalent meningococcal conjugate vaccine (MenACWY-CRM)
Arm/Group | MenACWY-CRM (A) | MenACWY-CRM (C) | MenACWY-CRM (W-135) | MenACWY-CRM (Y)
Number analyzed (Participants) | 23 | 23 | 23 | 23
titer | 54 [34 to 85] | 42 [27 to 66] | 90 [58 to 139] | 36 [16 to 81]

4. Primary Outcome: Percentage of Participants With Serum Bactericidal Activity of the Meningococcal ACWY Vaccine at One Month After Vaccination
Description: as for outcome 2
Time Frame: One month after vaccinations
Population: The analysis was done on the per protocol population.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MenACWY-CRM (A) | MenACWY-CRM (C) | MenACWY-CRM (W-135) | MenACWY-CRM (Y)
Number analyzed (Participants) | 23 | 23 | 23 | 23
percentage
  titers ≥ 4 | 96 [78 to 100] | 100 [85 to 100] | 100 [85 to 100] | 83 [61 to 95]
  titers ≥8 | 96 [78 to 100] | 96 [78 to 100] | 100 [85 to 100] | 83 [61 to 95]

5. Primary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions Post Vaccination.
Description: The number of subjects who reported solicited reactions after the administration of the Meningococcal B vaccine at a 0, 2, 6-month schedule and the administration of the Meningococcal A, C, W, and Y vaccine at month 7.
Time Frame: One month after vaccinations
Population: The analysis was done on the per protocol population.
Measure: Number; unit: participants
Groups:
- 4CMenB (Post Dose 1): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. We report Numbers (%) of Subjects with Local and Systemic Reactions as indicators of Reactogenicity, by Vaccination post dose 1
- 4CMenB (Post Dose 2): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. We report Numbers (%) of Subjects with Local and Systemic Reactions as indicators of Reactogenicity, by Vaccination post dose 2.
- 4CMenB (Post Dose 3): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. We report Numbers (%) of Subjects with Local and Systemic Reactions as indicators of Reactogenicity, by Vaccination post dose 3.
- Men ACWY-CRM (One Dose): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB. We report Numbers (%) of Subjects with Local and Systemic Reactions as indicators of Reactogenicity, by Vaccination post one dose of Men ACWY vaccine.
Arm/Group | 4CMenB (Post Dose 1) | 4CMenB (Post Dose 2) | 4CMenB (Post Dose 3) | Men ACWY-CRM (One Dose)
Number analyzed (Participants) | 53 | 52 | 50 | 41
participants
  Injection pain (any) | 52 | 50 | 50 | 10
  Injection pain (severe) | 8 | 7 | 9 | 0
  Erythema (any) | 22 | 23 | 28 | 9
  Erythema (severe) | 0 | 0 | 0 | 0
  Induration (any) | 23 | 24 | 29 | 5
  Induration (severe) | 0 | 0 | 0 | 0
  Nausea (any) | 7 | 5 | 9 | 4
  Nausea (severe) | 2 | 0 | 0 | 0
  Malaise (any) | 16 | 17 | 26 | 11
  Malaise (severe) | 3 | 1 | 2 | 1
  Myalgia (any) | 15 | 19 | 24 | 5
  Myalgia (severe) | 3 | 3 | 7 | 1
  Arthralgia (any) | 10 | 12 | 20 | 6
  Arthralgia (severe) | 0 | 0 | 3 | 0
  Headache (any) | 15 | 13 | 21 | 9
  Headache (severe) | 2 | 0 | 0 | 1
  Fever (≥ 38°C) | 2 | 1 | 0 | 2
  Stayed home | 5 | 4 | 5 | 2
  Analgesic, antipyretic medicine used | 10 | 7 | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (8 months).
Description: Adverse events categorized as systematic assessment is defined as solicited adverse events.
Groups:
- 4CMenB (1st Vaccination): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB.
  Post dose 1.
- 4CMenB (2nd Vaccination): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB.
  Post dose 2.
- 4CMenB (3rd Vaccination): All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB.
  Post dose 3.
- Men ACWY-CRM: All participants were administered three doses of 4CMenB (0,2,6 months) and all were administered a single dose of MenACWY-CRM 1 month after the third dose of 4CMenB.
  Post dose 1 MenACWY.
Arm/Group | 4CMenB (1st Vaccination) | 4CMenB (2nd Vaccination) | 4CMenB (3rd Vaccination) | Men ACWY-CRM
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/50 | 0/41
Other Adverse Events (participants affected / at risk) | 52/53 | 51/52 | 50/50 | 19/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4CMenB (1st Vaccination) (N=53) | 4CMenB (2nd Vaccination) (N=52) | 4CMenB (3rd Vaccination) (N=50) | Men ACWY-CRM (N=41)
Injection site pain (General disorders) | 52 | 50 | 50 | 10 — After first vaccination
Injection site induration (General disorders) | 23 | 24 | 29 | 5
Injection site erythema (General disorders) | 22 | 23 | 28 | 9
Headache (Nervous system disorders) | 16 | 13 | 21 | 9
Malaise (General disorders) | 16 | 17 | 26 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 19 | 24 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 12 | 20 | 6
Nausea (Gastrointestinal disorders) | 7 | 5 | 9 | 4
Pyrexia (General disorders) | 3 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less